CLINICAL TRIAL: NCT03347344
Title: Multicenter, Randomized, Double Blind, Placebo Controlled Clinical Trial With Riluzole in Spinocerebellar Ataxia Type 2
Brief Title: Clinical Trial With Riluzole in Spinocerebellar Ataxia Type 2 (ATRIL)
Acronym: ATRIL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P160927J; 2017-001481-23 (EudraCT Number)
Record Dates: First submitted 2017-09-21; First posted 2017-11-20 (Actual); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Spinocerebellar Ataxia Type 2
Keywords: Spinocerebellar ataxia-SCA2; SARA (Scale for the Assessment and Rating of Ataxia) score; Riluzole (Rilutek)
MeSH Terms: conditions — Spinocerebellar Ataxias | interventions — Riluzole

STUDY DESIGN:
Intervention Model Description: Multi-centric, double-blind randomized, two-arm controlled study (one group with 50 mg riluzole twice a day versus one group with placebo), during one year
Who Masked: Participant, Care Provider, Investigator
Masking Description: Treatments will be presented in numbered boxes, labeled for this study according to the Good Manufacturing Practices by the General Agency of Equipment and Health Products (AGEPS).
  Each numbered box will consist of 6 months of treatment: 20 blister packs of 20 active or placebo tablets
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RILUZOLE (Experimental): Riluzole PMCS 50 mg is presented as a round, biconvex, 8 mm diameter nearly white film-coated tablet. The tablets will be held under a blister of 20 tablets.
  Interventions: Drug: Riluzole
- PLACEBO (Placebo Comparator): The placebo PMCS 50 mg is presented as a round, biconvex, 8 mm diameter nearly white film-coated tablet matching the appearance of the Riluzole used in this study
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riluzole — 50 mg will be administered (per os) twice a day
  Arms: RILUZOLE
Drug: Placebo — 50 mg will be administered (per os) twice a day
  Arms: PLACEBO

SUMMARY:
ATRIL is a multi-centric, double-blind randomized, two-arm controlled study. 42 SpinoCerebellar Ataxia type 2 (SCA2) patients, both gender, at least 18 years of age will be included.

Riluzole 50 mg will be administered (per os) twice a day, versus one group with placebo for 12 months.

Riluzole (Rilutek®) is a benzothiazole drug, market approved, for Amyotrophic Lateral Sclerosis (ALS). It delays the onset of ventilator-dependence or tracheostomy in selected patients and may increase survival.

Scale for the Assessment and Rating of Ataxia (SARA) will be used at M0, M6 and M12. To assess primary criterion, the percentage of patients with a decrease of at least 1 point of the SARA score between the inclusion visit, and Visit 3 (Months 12) will be calculated.

DETAILED DESCRIPTION:
Inherited cerebellar ataxias are genetically heterogeneous neurological disorders. They are characterized by ataxic gait and cerebellar dysarthria that progresses over time with loss of ambulation and speech. The mutations by expansions of CAG triplets in the genes ATXN1 (SCA1), ATXN 2 (SCA2), 3 (SCA3), CACNA1A (SCA6), ATXN 7 (SCA7), and TBP (SCA17) are responsible for 50% of hereditary forms There is no curative or preventive treatment. This phase III study is a multi-centric, double-blind randomized, two-arm controlled study (one group with 50 mg Riluzole twice a day versus one group with placebo), to measure the efficacy of treatment with riluzole in SCA2 patients during 12 months. Amelioration is defined by a 1 point decrease of the SARA score.

ELIGIBILITY:
Inclusion Criteria:

* Genetically diagnosed SCA2 (CAG triplet in ATXN2 ≥ 33)
* At least 18 years of age
* Signature of informed consent
* Covered by social security
* SARA score ≥ 5 and ≤ 26
* Age at onset ≤ 50 years old

Exclusion Criteria:

* Treated with riluzole prior to the study
* Hepatotoxic medication
* Hypersensitivity to the active substance or to any of the excipients
* Serious systemic illnesses or conditions known for enhancing the side effects of riluzole
* Contraindications for MRI examination
* Participation in another therapeutic trial (3 months exclusion period)
* Pregnancy or breastfeeding
* Non abstinence or absence of effective contraception for women
* Inability to understand information about the protocol
* Persons deprived of their liberty by judicial or administrative decision
* Adult subject under legal protection or unable to consent
* Other ataxic syndromes than SCA2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2020-12-14 (Actual); Study Completion 2020-12-14 (Actual)

PRIMARY OUTCOMES:
Change in Ataxia symptoms (Scale for the Assessment and Rating of Ataxia (SARA)) | at 12 months.
  To compare the proportion of patients with Scale for the Assessment and Rating of Ataxia (SARA) improvement (decrease) of at least one point from baseline to 12 months

SECONDARY OUTCOMES:
Change in Ataxia symptoms (Composite Cerebellar Functional Severity (CCFS) score) | at 12 months
  To compare the difference of the CCFS score (Composite Cerebellar Functional Severity Score) from baseline at 12 months. A decrease is expected in the intervention group.
Change in extracerebellar symptoms (Inventory of Non-Ataxia Signs (INAS)) | at 12 months
  To compare the difference of the extracerebellar symptoms (INAS, Inventory of Non-Ataxia Signs) by showing decrease in the INAS count from baseline at 12 months
12 months survival | at 12 months
  To compare survival of the patients between the two treatment groups at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: DURR Alexandra, PU-PH, Principal Investigator — ASSISTANCE PUBLIQUE HÖPITAUX DE PARIS
Locations (1):
- Durr, Paris, France

REFERENCES:
- [Derived] Coarelli G, Heinzmann A, Ewenczyk C, Fischer C, Chupin M, Monin ML, Hurmic H, Calvas F, Calvas P, Goizet C, Thobois S, Anheim M, Nguyen K, Devos D, Verny C, Ricigliano VAG, Mangin JF, Brice A, Tezenas du Montcel S, Durr A. Safety and efficacy of riluzole in spinocerebellar ataxia type 2 in France (ATRIL): a multicentre, randomised, double-blind, placebo-controlled trial. Lancet Neurol. 2022 Mar;21(3):225-233. doi: 10.1016/S1474-4422(21)00457-9. Epub 2022 Jan 18. PMID 35063116